CLINICAL TRIAL: NCT02379598
Title: Effect of Therapy With Aminoacid Based Formula Versus Hydrolyzed Whey Proteins in Children With Cow's Milk Allergy
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Other Study IDs: 202/2011
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Amino acid based formula
  Interventions: Dietary Supplement: Aminoacid based formula
- Whey protein formula
  Interventions: Dietary Supplement: Hydrolyzed whey formula

INTERVENTIONS:
Dietary Supplement: Aminoacid based formula — Formula based on aminoacid
  Groups: Amino acid based formula
Dietary Supplement: Hydrolyzed whey formula — Formula based on hydrolyzed whey protein
  Groups: Whey protein formula

SUMMARY:
Cow's milk allergy is an immunologically mediated adverse reaction to milk proteins. In industrialized countries there is an incidence of 2-3% in children younger than 2 years. Cow's milk allergy may present with different clinical pictures and symptoms often nonspecific. Among the most common are certainly food refusal and failure to thrive until frameworks frank malnutrition. It was also noted that the cow's milk allergy can have a negative impact on the quality of life of the patient and his family.

The treatment of this condition provides the setting of a diet that is free of the allergen to the base of the adverse reaction.

There are some types of formulas for the treatment of this condition. The formulas based on amino acids are currently used in all cases non-responsive to treatment with the above formulas or in all those characterized by severe allergic reactions. Being made from amino acids such formulas are by definition non-allergenic. They have also proven to ensure a rapid resolution of symptoms favoring a resumption of growth, nutritional status, as well as lead to a rapid improvement in the quality of life of the patient and his family. However, the studies currently available to us concerning the effects of nutritional formulas based on amino acids affect short observation periods (usually less than 6 months) and were directed to a comparison only with hydrolysates of whey protein or casein and not with healthy subjects. To date thus lack consistent data on the nutritional effects in the medium to long term.

ELIGIBILITY:
Inclusion Criteria:

* subjects with diagnosis of cow's milk allergy

Exclusion Criteria:

* age <5 months
* age >12 months
* other concomitant chronic diseases
* malformations
* other food allergies

Ages: 5 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with a sure diagnosis of cow's milk allergy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
change of z-score weight at 12 months | after 12 months of intervention

SECONDARY OUTCOMES:
change of body mass index at 12 months | after 12 months of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- university of naples federico II, Naples, Naples, Italy

REFERENCES:
- [Derived] Canani RB, Nocerino R, Frediani T, Lucarelli S, Di Scala C, Varin E, Leone L, Muraro A, Agostoni C. Amino Acid-based Formula in Cow's Milk Allergy: Long-term Effects on Body Growth and Protein Metabolism. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):632-638. doi: 10.1097/MPG.0000000000001337. PMID 27437928